CLINICAL TRIAL: NCT06272747
Title: A Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetics of XH-S003 After Single Ascending Doses, Multiple Ascending Doses and Evaluation of Food Effects in Healthy Volunteers
Brief Title: Study of XH-S003 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: S-INFINITY Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-S003-I-101
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: A (XH-S003) (Experimental): Participants will receive XH-S003 once or twice daily on scheduled day(s)
  Interventions: Drug: XH-S003
- Placebo Comparator: B (Placebo) (Placebo Comparator): Participants will receive matching placebo once daily on scheduled day(s)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XH-S003 — IP: XH-S003 Dose: 25 mg, 100 mg Dose Formulation: Capsule Route of Administration: Oral
  Arms: Experimental: A (XH-S003)
Drug: Placebo — Dose: 25 mg, 100 mg Dose Formulation: Capsule Route of Administration: Oral
  Arms: Placebo Comparator: B (Placebo)

SUMMARY:
The purpose of the study is to assess the safety, tolerability and pharmacokinetics of XH-S003 in healthy volunteers under SAD (Single ascending dose) and MAD (Multiple ascending dose) studies. In addition, this study evaluates the food effects of XH-S003.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 to ≤ 55 years old.
2. BMI between ≥ 19.0 and ≤ 30.0 kg/m2 at Screening, and weight between ≥ 50 kg and ≤ 120.0kg for male, weight ≥ 45 kg and ≤ 120.0kg for female.
3. Able and willing to comply with the study procedure and the restriction specified in the protocol.
4. Provision of signed and dated written informed consent prior to any study specific procedures.
5. Female subjects of childbearing potential must have a negative serum pregnancy test result at screening and a negative pregnancy test result at baseline, and agree to use one of the acceptable methods of contraception listed below during the study (from the time of signing the informed consent until one month after the end of study [EOS] or early termination visit evaluation [ET]):

   * The subject's male partner has undergone documented vasectomy with documentation of azoospermia (male sterilization).
   * A documented placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * Consistent use of the same oral contraceptives for at least 3 months before screening, injectable progesterone, subdermal implants, or the use of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps], which present no effect on IP at the discretion of investigator).
   * Documented tubal ligation (female sterilization).
   * True abstinence: when this is in line with the preferred and usual lifestyle of the subject, including female subjects with same sex partners. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Abstinent subjects must agree to use one of the above-mentioned contraceptive methods, if they start sexual relationships during the study.

Exclusion Criteria:

1. Subjects with a history of allergies to similar ingredients of the study drug or any ingredient in the study drug, or vaccine component; subjects with a history of severe allergic or anaphylactic reactions at the discretion of PI. Subjects with one of the conditions (including, but not limited to):

   * Subjects with history of eczema within 3 years.
   * Subjects with asthma except for resolved childhood asthma.
   * Subjects with clinical syndromes of urticaria at screening or baseline.
2. Subjects whose abnormalities in past medical history are clinically significant or other clinical findings suggest the following clinically significant diseases at the discretion of the PI (including but not limited to gastrointestinal, renal, hepatic, neurological, hematologic, endocrine, pulmonary, psychiatric, or cardiovascular and cerebrovascular diseases, which are deemed as clinically significant by PI).
3. Abnormal liver function tests at screening, defined as alanine aminotransferase (ALT) or aspartate transaminase (AST) > 1.5x upper limit of normal (ULN), and bilirubin >1.5x ULN (isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) that are considered by the PI to be clinically significant. Repeat tests are permitted at investigator discretion.
4. Abnormal ECG findings at Screening or Day -1 (eg, repeated demonstration of a QTc interval > 450 ms [male] or > 470 ms [female] corrected by Fridericia's formula [QTcF] or Bazett's formula [QTcB]; heart rate [HR] is out of normal range 45-100 bmp; PR is out of normal range 120 -220 msec; QRS is out of normal range <120msec) that are considered by the PI or designee to be clinically significant. Repeat tests are permitted at investigator discretion.
5. Subjects with clinically significant infection (e.g., requiring hospitalization or parenteral antimicrobial therapy) within 2 months before screening or active systemic bacterial, viral, or fungal infection or fever with ear temperature > 37.7℃ within 2 weeks before screening at the discretion of the PI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Part A: Approximately 1~2 weeks
  Safety and tolerability evaluation: All participants were observed for any adverse events that occurred during the clinical study, including abnormalities in clinical symptoms and vital signs, physical examination, laboratory examination, and 12-lead electrocardiogram, and were determined to be associated with the investigational drug.
Number of participants with adverse events (AEs) | Part B: Approximately 3~4weeks
  Safety and tolerability evaluation: All participants were observed for any adverse events that occurred during the clinical study, including abnormalities in clinical symptoms and vital signs, physical examination, laboratory examination, and 12-lead electrocardiogram, and were determined to be associated with the investigational drug.
Number of participants with adverse events (AEs) | Part C: Approximately 3~4weeks
  Safety and tolerability evaluation: All participants were observed for any adverse events that occurred during the clinical study, including abnormalities in clinical symptoms and vital signs, physical examination, laboratory examination, and 12-lead electrocardiogram, and were determined to be associated with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital,Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No